CLINICAL TRIAL: NCT00521326
Title: Diagnosis and Characterization of Coronary Artery Stenosis by Transthoracic Doppler Ultrasound
Brief Title: Diagnosis and Characterization of Coronary Artery Stenosis by Doppler Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: DOP01
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-03

CONDITIONS: Coronary Stenosis
Keywords: doppler; coronary stenosis; non-invasive testing; A prospective study of a new diagnostic method.; Study consists of a transthoracic doppler of LAD.; Doppler to be performed prior to coronary angiography.; F/U doppler examination for those who undergo PCI.; Doppler results will be compared with coronary angiography.
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with an acute coronary syndrome that are candidates for coronary angiography. Doppler results will be compared to angiographic findings.

SUMMARY:
The purpose of this study is to evaluate the feasibility of acquisition of coronary blood flow velocity signals over the whole length of the LAD with transthoracic pulsed Doppler, and to evaluate the diagnostic power of the transthoracic Doppler analysis package for detecting and estimating the degree of coronary artery stenosis. Finally we hope to optimize the currently available analysis package on the basis of the comparison of the Doppler with the angiographic stenosis results and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically suspected of having significant coronary artery stenosis.
* Patients with CAD.
* Patients who are scheduled to undergo coronary angiography.
* Signed informed consent.

Exclusion Criteria:

* Patients with arrhythmia / irregular pulse
* Patients with unstable conditions: unstable angina, uncontrolled CHF
* Patients with COPD
* Any physical or medical disability that prevent lying in supine position
* Patients with chest wall deformity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Simcha R Meisel, MD, MSc, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Coronary Care Unit, Heart Institute, Hille Yaffe Medical Center, Hadera, Israel